CLINICAL TRIAL: NCT04188496
Title: The Effects of Thoracic Joint Mobilization on Pulmonary Functions of Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shehla Gul (Individual)
Responsible Party: Sponsor-Investigator, Shehla Gul, Principal Investigator, Gul, Shehla
Organization: Gul, Shehla (Individual)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU Shehla Gul
Record Dates: First submitted 2019-08-26; First posted 2019-12-06 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Stroke
Keywords: Pulmonary Functions; Stroke
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PULMONARY FUNCTION TEST (PFT) GROUP (Experimental): Thoracic joint Mobilization was applied on Experimental group.
  Thoracic Flexion:
  Patient sits on the treatment table with arms across the chest and hands on opposite shoulders. Stand facing the patient's left side.
  Thoracic Extension:
  Performed by asking sits on a treatment chair with arms folded across the chest and hands on opposite shoulders.
  Thoracic Segment Rotation:
  Performed by asking the patient to lie on left side. Place a pillow under patient's waist to assist left side bending. Position the patient's arms are folded across the chest with hands on opposite shoulders to stabilize the shoulder girdle and minimize movement there.
  Interventions: Other: Pulmonary Function Test group
- Control Group (Other): received conventional Chest physiotherapy Techniques for 30 minutes (including deep breathing, diaphragmatic breathing exercises, Self-stretching exercises for accessory respiratory muscles, Respiratory Resistance training by incentive spirometer) followed by 10 min rest.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Pulmonary Function Test group — The interventional group received the same conventional Chest physiotherapy Techniques for 30 minutes followed by 10 minutes rest. The patients then received additional 15 minutes protocol of thoracic joint mobilization
  Arms: PULMONARY FUNCTION TEST (PFT) GROUP
Other: Control Group — received conventional Chest physiotherapy Techniques for 30 minutes (including deep breathing, diaphragmatic breathing exercises, Self-stretching exercises for accessory respiratory muscles, Respiratory Resistance training by incentive spirometer) followed by 10 min rest.
  Arms: Control Group

SUMMARY:
Stroke a neurological disorder leads to long term disability and decline in overall quality of life. Pulmonary Functions are usually impaired in individuals with stroke. The common findings associated with pulmonary functions in Stroke patients are Decreased lung volumes, decreased pulmonary perfusion and vital capacity and altered chest wall excursion. For stroke patients, general rehabilitation programs, only aims towards their functional recovery of the body. The main focus of this study was to integrate intervention and implement them in rehabilitation programs that are related to respiration are more effective for improving functional activities.in stroke patients. The study was carried out to determine the effects of thoracic Joint Mobilization on Pulmonary Functions of patients with stroke.

DETAILED DESCRIPTION:
INTRODUCTION Stroke is defined as sudden neurological deficit due to an abnormality in cerebral blood flow, with sign and symptoms lasting for more than 24 hours. Strokes can be grouped into two fundamental classification according to the American Stroke Association (ASA), first is ischemic (87%) and the second is Hemorrhagic (13%). In epidemiological and genetic studies a stroke subtype classification is useful indicator in our clinical practice. Many serious physical and cognitive deficits results due to injury to the brain tissue. Depending upon the region of the brain that is involved and amount of damage, a person can recovers from stroke.

Stroke is associated with many primary and secondary complications. Here mentioned some primary complications. Sensation, Pain, Visual changes, Motor Function, Weakness, Alternation in Tone, Abnormal Reflexes, Altered Coordination, Altered Postural control and Balance. The main Indirect or secondary complications are Musculoskeletal Complications, Neurological Complications, Cardiovascular Complications, Pulmonary Complications, and Integumentary Complications.

Pulmonary Functions are usually impaired in individuals with stroke. The common findings associated with pulmonary functions in Stroke patients are Decreased lung volumes, decreased pulmonary perfusion and vital capacity and altered chest wall excursion. Individuals with stroke are, associated with dysphagia which leads to dehydration and compromised nutrition. Dysphagia has been related with enlarged risk of pulmonary difficulties and also death. According to research evidence primary findings of dysphagia in patients having acute stroke significantly decreases complications. It also decreases the length of hospital stay and overall health expenditure.

Dysphagia further leads to Aspiration. Aspiration, is penetration of food, liquid, saliva or gastric reflux into the airways. It usually occurs in acute phase of recovery or during swallowing. Aspiration is an important complication and can leads to aspiration pneumonia if left untreated, death can occur.

Impaired Pulmonary functions limits physical activities as well. Because the decreased respiratory output is accompanied by increased oxygen demands required during altered movement patterns in stroke. Furthermore people with stroke usually undergo irregular breathing because of damage to the respiratory muscles (such as Diaphragm).

Due to paralyzed respiratory muscles lungs and thorax cannot be sufficiently dilated. If this condition persists the thoracic tissues may become shortened and thoracic muscles undergo fibrosis to reduce the compliance of thorax. This leads to various complications like atelectasis, changes in muscles forces, which directly or indirectly obstruct the performance of daily living activities, and asymmetrical postures or movement foam, which may hamper the stability of motion there by.

In stroke patients the respiratory functions are affected both directly and indirectly by the cardiopulmonary performance because they experience a deterioration in cardiovascular functioning and pulse rate. This disturbs the oxygen delivery and decline in the activity of the chest wall on the paralyzed side and its electrical activities. The changes in breathing mechanism and respiratory efficiency reflects about the extent of loss in the activity of chest wall, loss of symmetry and the extent of muscular paralysis of stroke patients. To correct above mentioned difficulties it is significant to have expansion of chest wall, to improve lung ventilation and to have suitable volume and capacities of lungs.

As mentioned above stroke is accompanied by many secondary complications due to nervous system and musculoskeletal system insufficiencies related through brain impairments. Amongst many problems pulmonary disorders are further, strictly associated to life, difficulties with respiration and swallowing as well as language.

Direct restrictive impairments accompanied due to non-utilization of paralyzed muscles and their trouble with movement elicits a secondarily decrease in cardiopulmonary functioning. Due to this, non-symmetric trunk encourages insufficient energy use related to gait, causing reduction in exercise endurance. Patients having hemiplegia due to stroke experiences deviated movement in posture, abnormal movement of trunk and motor control.

Now a day's people preserve static posture for long periods due to which occurrence of cervical lordosis along with thoracic and lumbar kyphosis is growing day by day. Due to an inclination in thoracic kyphosis, restriction in expansion of chest and respiratory weakness of muscles occurs, thus decreasing lungs capacity and size of the thoracic cavity and distorting vertebral column arrangement.

Our study focuses on the effects of thoracic joints mobilization and its effects on enhancing the pulmonary functions in stroke patients. Generally Rehabilitation programs target towards functional recovery of body. They neglect enhancement of cardiopulmonary system functioning. If investigator incorporate interventions related to respiration along with functional recovery, it possibly be additionally effective in stroke patients for enhancing functional doings such as gait.

Many studies shows the effects of mobilization and its effects on pulmonary function. A study on The Immediate Effect of Chest Mobilization Technique on Chest Expansion in Patients of COPD with Restrictive Impairment. This study concluded that mobilization of rib cage joints improve ribcage mobility and reduced obstructive lung disease. Chest wall mobilization also improves the mobility of chest wall, reduces respiratory rate, increases tidal volume, improves ventilation, reduces dyspnea, decreases work of breathing and facilitate relaxation.

Another study focuses on, the effect of thoracic region self-mobilization on chest expansion and pulmonary function. The purpose of this study was to find out the effects of thoracic region self-mobilization on chest expansion and pulmonary function in healthy adults. The outcome measures included in this study were to measure chest expansion during breathing, pulmonary functions, and expected pulmonary functions. There was no noteworthy change in pulmonary functions among intervention and control group. There was a noteworthy change in chest expansion between intervention and control group. Hence concluded that thoracic region self-mobilization is helpful for improving chest expansion in healthy adults.

Our study focuses on the effects of thoracic joints mobilization and its effects on pulmonary functions in stroke patients. Generally Rehabilitation programs target towards functional recovery of body. They neglect enhancement of cardiopulmonary system functioning. If investigator incorporate interventions related to respiration along with functional recovery, it possibly be additionally effective in stroke patients for enhancing functional doings such as gait.

ELIGIBILITY:
Inclusion Criteria:

* A sample of 26 patients with stroke without any history of recent pulmonary involvement
* Diagnosed with stroke by computed tomography (CT) or magnetic resonance imaging (MRI), with disease duration of at least six months after the onset of stoke.
* Score 24 points or higher on MMSE to ensure that they able to understand and follows the researcher's order.

Exclusion Criteria:

* The subjects having any recent surgery,
* unstable blood pressure and
* having acute infections were excluded from the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
Forced expiratory Volume in one sec (FEV1) | 6 months
  Pulmonary Functions: Forced expiratory Volume in one sec (FEV1) was measured in litre/sec through digital spirometer
Forced vital capacity (FVC) | 6 months
  Pulmonary Functions: Forced vital capacity (FVC) was measured in litre through digital spirometer

CONTACTS AND LOCATIONS:
Locations (1):
- Shehla Gul, Attock, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Susuan B O'Sullivan TJS. Physical Rehabilitation and Medicine. 5 th Edition ed.
- [Background] [updated 9/24/14]. Available from: http://www.strokeeducation.info/types/index.htm.
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Jang SH, Bang HS. Effect of thoracic and cervical joint mobilization on pulmonary function in stroke patients. J Phys Ther Sci. 2016 Jan;28(1):257-60. doi: 10.1589/jpts.28.257. Epub 2016 Jan 30. PMID 26957769
- [Background] Seo K, Hwan PS, Park K. The effects of inspiratory diaphragm breathing exercise and expiratory pursed-lip breathing exercise on chronic stroke patients' respiratory muscle activation. J Phys Ther Sci. 2017 Mar;29(3):465-469. doi: 10.1589/jpts.29.465. Epub 2017 Mar 22. PMID 28356632
- [Background] Han JM, Kim H, Koo JP, Seo KC. Effects of respiratory muscle activity in stroke patients after feedback breathing exercise. Journal of International Academy of Physical Therapy Research. 2013;4(2):552-6.
- [Background] Amarenco P, Bogousslavsky J, Caplan LR, Donnan GA, Hennerici MG. Classification of stroke subtypes. Cerebrovasc Dis. 2009;27(5):493-501. doi: 10.1159/000210432. Epub 2009 Apr 3. PMID 19342825
- [Background] Lanini B, Bianchi R, Romagnoli I, Coli C, Binazzi B, Gigliotti F, Pizzi A, Grippo A, Scano G. Chest wall kinematics in patients with hemiplegia. Am J Respir Crit Care Med. 2003 Jul 1;168(1):109-13. doi: 10.1164/rccm.200207-745OC. Epub 2003 Apr 24. PMID 12714347
- [Background] Jung JH, Moon DC. The effect of thoracic region self-mobilization on chest expansion and pulmonary function. J Phys Ther Sci. 2015 Sep;27(9):2779-81. doi: 10.1589/jpts.27.2779. Epub 2015 Sep 30. PMID 26504292
- [Background] Song GB, Park EC. Effects of chest resistance exercise and chest expansion exercise on stroke patients' respiratory function and trunk control ability. J Phys Ther Sci. 2015 Jun;27(6):1655-8. doi: 10.1589/jpts.27.1655. Epub 2015 Jun 30. PMID 26180292
- [Background] Colby CKaLA. Therapeutic Exercise Foundations and Techniques. 5th ed.
- [Background] Kim J, Park JH, Yim J. Effects of respiratory muscle and endurance training using an individualized training device on the pulmonary function and exercise capacity in stroke patients. Med Sci Monit. 2014 Dec 5;20:2543-9. doi: 10.12659/MSM.891112. PMID 25488849
- [Background] Mohan V, Aziz KB, Kamaruddin K, Leonard JH, Das S, Jagannathan MG. Effect of intercostal stretch on pulmonary function parameters among healthy males. EXCLI J. 2012 Jun 15;11:284-90. eCollection 2012. PMID 27418905
- [Background] Hwangbo PN, Hwangbo G, Park J, Lee S. The Effect of Thoracic Joint Mobilization and Self-stretching Exercise on Pulmonary Functions of Patients with Chronic Neck Pain. J Phys Ther Sci. 2014 Nov;26(11):1783-6. doi: 10.1589/jpts.26.1783. Epub 2014 Nov 13. PMID 25435700